CLINICAL TRIAL: NCT00012493
Title: Cardiac Vulnerability in Potentially Susceptible Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 9825-CP-001
Record Dates: First submitted 2001-03-09; First posted 2001-03-12 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Heart Disease
Keywords: Cardiac event; Heart disease; Particulate Matter
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This project is part of a program project directed toward assessing cardiac effects of particulate and other ambient air pollutants. In this project patient who have recently suffered a cardiac event are being monitored with cardiac monitors for 24 hours up to 4 times during the year following their cardiac event. Similarly a second group of patients with moderate to severe heart failure will undergo similar cardiac monitoring for 24 hours, twice a week separated by 3 months. In both sets of patients home indoor pollution measures will be continuously made and used to correlate with measures of heart rate variability.

DETAILED DESCRIPTION:
Approximately 50 patients in each group will be studied. In addition to cardiac monitoring for 24 hours at each session, overnight respiratory pattern and oxygen saturation will be monitored in both groups. The exposure monitoring will include both particle mass of PM2.5 along with detailed assessment to determine that portion of the particulate exposure from outdoor vs. indoor sources.

ELIGIBILITY:
For the cardiac event cases patients are selected from the Brigham and Women's Hospital cardiac services at the time of discharge, aged 45-74, having suffered a cardiac event resulting in either an infarct or need for a cardiac procedure (angioplasty, stint, etc). For the CHF patients they are selected from the BWH cardiac clinics where they have been identified and classified as stage 3 or 4 CHF. For both groups residence requirements are that they reside within the Greater Boston Area as defined by an outer ring road (Route 495) and are willing to be visited at home and have the exposure assessment equipment set up in their home as well as be monitored personally.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1999-10; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Frank E Speizer, MD, Principal Investigator — Environmental Epidemiology Program, Department of Environmental Health, Harvard School of Public Health
Locations (1):
- Brigham and Womens Hospital, Boston, Massachusetts, United States